CLINICAL TRIAL: NCT05936229
Title: Phase 1/2 Study to Evaluate the Safety, Feasibility, and Efficacy of FP-1201 (Intravenous Interferon-Beta-1a) to Prevent Toxicities After CD19-Directed CAR T-Cell Therapy
Brief Title: Interferon-Beta-1a (FP-1201) to Prevent Toxicities After CD19-Directed CAR T-Cell Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed before opening to accrual, no participants enrolled
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1123521; NCI-2023-04888 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20021 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-05

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Recurrent B-Cell Non-Hodgkin Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory B-Cell Non-Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Mantle-Cell | interventions — Interferon beta-1a; X-Rays; Phantoms, Imaging; Magnetic Resonance Spectroscopy; Spinal Puncture; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (interferon beta-1A [FP-1201]) (Experimental): Patients undergo leukapheresis prior to treatment and receive FP-1201 IV for 3 days every 24 hours from day -3 through day -1 or for 5 days every 24 hours from day -5 through day -1 or on day -5, day -3, and day -1. Patients may receive lymphodepletion chemotherapy with either cyclophosphamide IV and fludarabine IV on days -5, -4, -3 followed by axi-cel IV or brexu-cel IV on day 0 or fludarabine IV over 30 minutes on days -4, -3, and -2 and cyclophosphamide IV over 60 minutes on day -2 followed by brexu-cel IV on day 0. Patients undergo x-ray imaging and ECHO or MUGA during screening. Patients also undergo CT or PET/CT as well as LP for CSF collection and/or bone marrow aspiration and biopsy as clinically indicated during screening and follow-up. Patients undergo blood sample collection on study and during follow-up as well as a tissue biopsy during screening and follow-up.
  Interventions: Biological: Interferon Beta-1A; Procedure: X-Ray Imaging; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Lumbar Puncture; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection; Procedure: Biopsy

INTERVENTIONS:
Biological: Interferon Beta-1A — Given IV
  Other Names: 145258-61-3; Avonex; BG9418; Rebif; Recombinant interferon beta-1a
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; Computed Axial Tomography; Computerized axial tomography (procedure)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging; Pet Scan; Positron emission tomography (procedure); Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; spinal tap
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase I/II trial tests the safety and how well intravenous interferon-beta-1a (FP-1201) works in preventing toxicities after CD19-directed chimeric antigen receptor (CAR) T-cell therapy in patients with B-cell cancers that has come back after a period of improvement (recurrent) or that has not responded to previous treatment (refractory). Interferon beta-1a is in a class of medications called immunomodulators. It works by protecting the lining of blood vessels, and preventing brain inflammation. Giving FP-1201 may prevent cytokine release syndrome (CRS) and immune effector cell associated-neurotoxicity syndrome (ICANS) toxicities in patients receiving CD19 CAR T-cell therapy with recurrent or refractory B-cell malignancies.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of FP-1201.

Patients undergo leukapheresis prior to treatment and receive FP-1201 intravenously (IV) for 3 days every 24 hours from day -3 through day -1 or for 5 days every 24 hours from day -5 through day -1 or on day -5, day -3, and day -1. Patients may receive lymphodepletion chemotherapy with either cyclophosphamide IV and fludarabine IV on days -5, -4, -3 followed by axi-cel IV or brexu-cel IV on day 0 or fludarabine IV over 30 minutes on days -4, -3, and -2 and cyclophosphamide IV over 60 minutes on day -2 followed by brexu-cel IV on day 0. Patients undergo x-ray imaging and echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo computed tomography (CT) or positron emission tomography (PET)/CT as well as lumbar puncture (LP) for cerebral spinal fluid (CSF) collection and/or bone marrow aspiration and biopsy as clinically indicated during screening and follow-up. Patients undergo blood sample collection on study and during follow-up as well as a tissue biopsy during screening and follow-up.

After completion of study treatment, patients are followed up to 28 days and 90 days, then long-term for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Karnofsky performance status of >= 60%
* Participants eligible for treatment with axi-cel or brexu-cel
* Negative serum pregnancy test within 2 weeks of enrollment for women of childbearing potential, defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year
* Fertile male and female participants must be willing to use an effective contraceptive method before, during, and for at least 4 months after the last dose of FP-1201
* Ability to understand and provide informed consent

Exclusion Criteria:

* Known hypersensitivity to natural or recombinant interferon beta, albumin or any other component of the formulation
* Estimated creatinine clearance (Cockcroft and Gault) =< 60 mL/min
* Significant proteinuria defined as 2+ or 3+ proteinuria or urinary protein >= 1g/24h
* Severe hepatic dysfunction defined as group C of the National Cancer Institute Organ Dysfunction Working Group hepatic impairment criteria (total bilirubin > 3x upper limit of normal [ULN] with any aspartate aminotransferase [AST] or alanine transaminase [AL]T value), or AST or ALT > 3x ULN, unless due to malignancy or Gilbert's syndrome in the opinion of the principal investigator (PI) or designee
* Participants with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing, as clinically indicated. Those with an forced expiratory volume in the first second (FEV1) of < 50 % of predicted or diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected) < 40% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following:

  * New York Heart Association (NYHA) class III or IV congestive heart failure, clinically significant hypotension
  * Uncontrolled symptomatic coronary artery disease, or a documented ejection fraction of < 35%
* Uncontrolled serious and active infection
* Corticosteroid use (> 20mg/day of prednisone, or equivalent) within 7 days prior to first FP-1201 administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rates | Within 14 days after the last administration of interferon-beta-1a (FP-1201)
  Will be summarized in the DLT evaluable population. Final DLT rates at each dose level will be estimated by isotonic regression by applying the pooled adjacent violators algorithm. The target toxicity rate is 30%.
Incidence of adverse events (AEs) | From the first dose of FP-1201 through day 28 after chimeric antigen receptor (CAR) T-cell infusion
  Type, frequency, and severity of AEs according to the National Cancer Institutes Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Cytokine release syndrome (CRS) rates | From the time of CAR T-cell infusion through day 28 after CAR T-cell infusion or until resolution, whichever happens last
  Will be assessed by any grade and grade >= 3 by American Society for Transplantation and Cellular Therapy (ASTCT) criteria and will be summarized along the two-sided 95% Clopper-Pearson confidence interval (CI) based on the CRS and ICANS analysis set.
Immune effector cell associated-neurotoxicity syndrome (ICANS) rates | From the time of CAR T-cell infusion through day 28 after CAR T-cell infusion or until resolution, whichever happens last
  Will be assessed by any grade and grade >= 3 by ASTCT criteria and will be summarized along the two-sided 95% Clopper-Pearson CI based on the CRS and ICANS analysis set.
Cumulative corticosteroids dose | Within 28 days after CAR T-cell infusion
  Will be summarized using descriptive statistics (median, quantiles) based on the CRS and ICANS analysis set.
Overall response rate | 28 days after CAR T-cell infusion
  Will be assessed by the Lugano criteria for B-non-Hodgkin lymphoma (NHL) participants and National Comprehensive Cancer Network (NCCN) criteria for B- acute lymphoblastic leukemia (ALL) participants Will be summarized along with the two-sided Clopper-Pearson CI based on the anti-tumor response evaluable analysis set.
Complete response rate | 28 days after CAR T-cell infusion
  Will be assessed by the Lugano criteria for B-NHL participants and NCCN criteria for B-ALL participants Will be summarized along with the two-sided Clopper-Pearson CI based on the anti-tumor response evaluable analysis set.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Gauthier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No